CLINICAL TRIAL: NCT04211584
Title: Randomized Controlled Trial Comparison Between Traditional ENtry Point and Distal puncturE of RAdial Artery (TENDERA Trial)
Brief Title: The TENDERA Multicenter Clinical Trial
Acronym: TDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Endosurgery and Lithotripsy, Moscow, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEN-001/18
Record Dates: First submitted 2018-02-25; First posted 2019-12-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Artery; Thrombosis
Keywords: Transradial intervention,radial artery,anatomic snuffbox
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor is blinded regarding used access site (traditional radial or Snuffbox approach)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- forearm radial artery access (Active Comparator): traditional access (puncture and cannulation) in the forearm part of the radial artery will be made for further coronary interventions
  Interventions: Device: transradial interventions
- anatomic snuffbox access (Active Comparator): access in the snuffbox area of the wrist (puncture and cannulation) in the forearm part of the radial artery will be made for further coronary interventions
  Interventions: Device: transradial interventions

INTERVENTIONS:
Device: transradial interventions — percutaneous coronary interventions in stable patients - diagnostic and treatment

SUMMARY:
TENDERA is a multicenter randomized controlled trial to compare traditional entry point in the radial artery for TRI and distal puncture at the anatomical snuffbox area for transradial Interventions. The Investigators hypothesized that novel entry point in radial artery may lessen vascular access site complication rate and especially the radial artery late occlusion rate.

DETAILED DESCRIPTION:
the forearm access will be made using traditional technique what was well described previously in the literature. The novel puncture site is located in the snuffbox area distal to the traditional radial access point. Thanks to surrounded anatomical conditions in anatomical snuffbox area vascular access site complications may be lessened comparing to forearm radial access site.

ELIGIBILITY:
Inclusion Criteria:

age 18-75 primary radial artery puncture radial artery diameter >1,5mm by ultrasound stable coronary disease less than 6F sheath needed patient height >185cm

Exclusion Criteria:

ACS AMI critically ill patients previous TRI procedure Raynaud's disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 850 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2021-09-18 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Radial artery late occlusion | 1 year
  loss of pulse or absent of artery lumen by ultrasound examonation

SECONDARY OUTCOMES:
vascular access site related complications | 1 week, 3 months, 6 moths, 1 year
  hematomas >5cm, bleeding, false aneurism, arterio-venous fistula

CONTACTS AND LOCATIONS:
Overall Officials: Avtandil M Babunashvili, MD, Principal Investigator — Center of Endosurgery; Alexander Kaledin, MD, Principal Investigator — North West state University Saint Petersburg
Locations (1):
- Center of Endosurgery, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IV Q of 2021 after the end of the study
Access Criteria: IPD may be requested by interventional cardiologists or radiologists IPD information may be shared after a request from individual or academic organizations if some concern and questions will raised

REFERENCES:
- [Derived] Babunashvili AM, Pancholy S, Zulkarnaev AB, Kaledin AL, Kochanov IN, Korotkih AV, Kartashov DS, Babunashvili MA. Traditional Versus Distal Radial Access for Coronary Diagnostic and Revascularization Procedures: Final Results of the TENDERA Multicenter, Randomized Controlled Study. Catheter Cardiovasc Interv. 2024 Dec;104(7):1396-1405. doi: 10.1002/ccd.31271. Epub 2024 Oct 30. PMID 39474765